CLINICAL TRIAL: NCT00002127
Title: A Phase II, Parallel Group, Randomized, Placebo-Controlled Study of the Safety and Efficacy of Thalidomide in Reducing Weight Loss in Adults With HIV Wasting Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 230A; W-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: Acquired Immunodeficiency Syndrome; Cachexia; Thalidomide
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome; Acquired Immunodeficiency Syndrome; Cachexia | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
To evaluate the safety, antiviral and anti-TNF-alpha activity, and preliminary efficacy of thalidomide in reducing weight loss in patients with HIV wasting syndrome.

DETAILED DESCRIPTION:
Patients are randomized to receive either thalidomide at 1 of 2 doses or placebo for 8 weeks. Patients who respond may continue in double-blinded treatment for an additional 4 weeks; nonresponding patients may receive thalidomide for up to 4 weeks. Per amendment, patients may receive thalidomide for more than 12 weeks on a compassionate basis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Primary prophylaxis for opportunistic infections (if AFB blood culture negative).
* Chronic suppressive therapy (maintenance) for opportunistic infections OTHER THAN Mycobacterium avium Complex (MAC).

Patients must have:

* Documented HIV infection.
* Wasting syndrome.
* Negative blood PCR for acid-fast bacteria (AFB) or a negative AFB blood culture within 48 days prior to study entry.
* No active opportunistic infection requiring systemic therapy within 6 weeks prior to study entry.
* Life expectancy of at least 6 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Chronic diarrhea (five or more unformed stools per day).
* Peripheral neuropathy of grade 2 or worse.
* Requirement for tube feeding or intravenous feeding.
* Any disorder associated with moderate to severe edema (e.g., cirrhosis, nephrosis, congestive heart failure).
* Inability to ingest at least a maintenance diet based on present weight.
* Any condition that precludes study participation.
* Not under the care of a primary physician.

Concurrent Medication:

Excluded:

* Chronic suppressive therapy (maintenance) or secondary prophylaxis for Mycobacterium avium Complex (MAC) (suppressive therapy for other opportunistic infections is allowed).

Concurrent Treatment:

Excluded:

* Radiotherapy.

Patients with the following prior conditions are excluded:

* Any neoplasms other than non-medicated (i.e., not receiving systemic or intralesional chemotherapy) Kaposi's sarcoma within 1 month prior to study entry.
* Prior intolerance to thalidomide.

Prior Medication:

Excluded:

* ddC within 1 month prior to study entry.
* Acute systemic therapy for opportunistic infections within 6 weeks prior to study entry.
* Agents that are anabolic, catabolic, or immunomodulatory (including interferons, megestrol, dronabinol, oxandrolone, growth hormone, systemic corticosteroids, and pentoxifylline) within 30 days prior to study entry.

Prior Treatment:

Excluded:

* Radiotherapy within 6 weeks prior to study entry.

Required ONLY IF patient is on antiretroviral therapy:

* Stable regimen of AZT or ddI for at least 1 month prior to study entry. Active drug abuse within 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Marin County Specialty Clinic, Greenbrae, California
  - AIDS Community Research Consortium, Redwood City, California
  - UCSD Med Ctr - Owen Clinic, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Gottlieb Med Group, Sherman Oaks, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Rockefeller Univ, New York, New York
  - Thomas Jefferson Med College, Philadelphia, Pennsylvania
  - Advanced Research Management, Seattle, Washington

REFERENCES:
- [Background] Stirling D, Sherman M, Strauss S. Thalidomide. A surprising recovery. J Am Pharm Assoc (Wash). 1997 May-Jun;NS37(3):306-13. PMID 9170807